CLINICAL TRIAL: NCT00934206
Title: Pilot Study to Find Predictors of Individual Training Effectiveness in Preventive Exercise
Brief Title: Predictors of Individual Training Effectiveness in Preventive Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Anne Krieg M.D., Institute of Sports- and Preventive Medicine, Saarland University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01/2009
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-06

CONDITIONS: Primary Prevention
Keywords: Exercise; healthy subjects
MeSH Terms: conditions — Motor Activity | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Training (Experimental): One month of endurance training (running / walking at 60 % heart rate reserve for 45 min 4 times per week)
  Interventions: Behavioral: Endurance training

INTERVENTIONS:
Behavioral: Endurance training — running / walking at 60 % heart rate reserve 4 times per week for 4 weeks

SUMMARY:
Physical exercise elicits beneficial changes in the body. These concern physical performance but also improvements in virtually all known risk factors for cardiovascular disease. Yet, the extent of individual benefit differs considerably even within homogenous groups and the prediction of individual training effectiveness is not yet possible. This study aims to find predictors of individual training effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* age 35-60

Exclusion Criteria:

* Any medical condition requiring medication (except thyroid hormones)
* Other complaints that might interfere with exercise

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
correlation of possible predictors with training effects on cardiovascular risk factors | within study periode

SECONDARY OUTCOMES:
Correlation of possible predictors with improvements in physical performance | within study period

CONTACTS AND LOCATIONS:
Overall Officials: Anne Krieg, M.D., Principal Investigator — Institute of Sports- and Preventive Medicine, Saarland University
Locations (1):
- Institute of Sports- and Preventive Medicine, Saarland University, Saarbrücken, Saarland, Germany

REFERENCES:
- [Derived] Hecksteden A, Grutters T, Meyer T. Associations between acute and chronic effects of exercise on indicators of metabolic health: a pilot training trial. PLoS One. 2013 Nov 21;8(11):e81181. doi: 10.1371/journal.pone.0081181. eCollection 2013. PMID 24278393
- See also: Primary sponsor and study location — http://www.sportmedizin-saarbruecken.de